CLINICAL TRIAL: NCT05243576
Title: A Novel System for Quasi Real-Time Tracking of Neuromuscular Responses During Electrical Stimulation
Brief Title: A Novel System for Quasi Real-Time Tracking of Neuromuscular Responses During NMES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Collaborators: New Jersey Commission on Spinal Cord Research (Other)
Responsible Party: Principal Investigator, Rakesh Pilkar, Senior Research Scientist, Kessler Foundation
Other Study IDs: R-1103-20
Record Dates: First submitted 2022-02-07; First posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Spinal Cord Injuries; Incomplete Spinal Cord Injury
Keywords: Neuromuscular Electrical Stimulation; Electromyography; EMG-feedback; Spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- incomplete SCI: 1) Be motor incomplete; 2) Be AIS classified as C or D; 3) have a neurological level of injury from C6 - T6; 4) Have LEMS score > 10; 5) Have Modified Ashworth Scale ≤ 3 for spasticity.
  Additional - 1) Be able to tolerate electrical stimulation; 2) Be able and willing to comply with study requirements, procedures and verbal instructions; 3) Have been diagnosed with a spinal cord injury by a physician.
- complete SCI: 1) Be chronic (≥ 1-year post injury); 2) AIS classified as A or B motor-complete;
  Additional - 1) Be able to tolerate electrical stimulation; 2) Be able and willing to comply with study requirements, procedures and verbal instructions; 3) Have been diagnosed with a spinal cord injury by a physician.
- Able-bodied: 1) Be able and willing to tolerate electrical stimulation; 2) Be able and willing to comply with study requirements, procedures and verbal instructions.

SUMMARY:
Neuromuscular electrical stimulation (NMES) remains as one of the effective rehabilitation modalities for addressing recovery of neuromuscular function after a spinal cord injury (SCI). To achieve optimal effects, the NMES interventions that involve or promote voluntary efforts from SCI participants are preferred. However, these interventions are limited by the fact that the active monitoring of voluntary effort, particularly at the stimulated muscle level is unattainable. The objective of the proposed study is to develop SMARTq (Stimulated Muscle Assessment in Real-Time). This novel system will provide a quasi real-time assessment of intrinsic neuromuscular responses of a stimulated muscle during NMES. Specifically, the proposed system will consist of our novel algorithms interfaced with the EMG data acquisition hardware to process the EMG data recorded from a stimulated muscle in real-time during NMES. The term 'quasi' is used to account for the processing delay of approximately 1 to 2 seconds that may potentially occur. The proposed system will be developed and validated using the data collected from the able-bodied (AB) as well as individuals with incomplete SCI (iSCI). The applicability of the system will be evaluated on individuals with complete SCI (cSCI). Our central hypothesis is that the real-time tracking of neuromuscular responses during a train of NMES will provide valuable information on inherent neuromuscular changes, volitional participation, and neuromuscular recovery. The significance of the proposed study is that, if successful, it will deliver a highly novel system which can allow researchers and clinicians to - 1) evaluate the direct electrophysiological effects of varied combination of NMES on a stimulated muscle in real-time; 2) quantify, track and manipulate the levels of voluntary efforts or volitional drive 'on-fly' during NMES for extracting optimal benefits; 3) track the neuromuscular recovery of the stimulated muscle, particularly for cSCI populations, when any functional changes have not been observed yet; and 4) directly observe the neuromuscular fatigue derived from the electrophysiological data at the stimulated muscle. These are highly significant opportunities that can allow the clinicians and researchers to transform the current as well as future NMES interventions into highly effective training modalities as each intervention will be operated at an individual's neuromuscular level.

ELIGIBILITY:
Inclusion Criteria:

SCI generic criteria - 1) Be able to tolerate electrical stimulation; 2) Be able and willing to comply with study requirements, procedures and verbal instructions; 3) Have been diagnosed with a spinal cord injury by a physician.

Individuals with complete SCI. 1) Be chronic (≥ 1-year post injury); 2) AIS classified as A or B motor-complete;

Individuals with incomplete SCI. 1) Be motor incomplete; 2) Be AIS classified as C or D; 3) have a neurological level of injury from C6 - T6; 4) Have LEMS score > 10; 5) Have Modified Ashworth Scale ≤ 3 for spasticity.

Inclusion criteria for the able-bodied group. 1) Be able and willing to tolerate electrical stimulation; 2) Be able and willing to comply with study requirements, procedures and verbal instructions.

Exclusion Criteria:

Exclusion criteria for all participants. 1) Pregnancy at time of study; 2) History of femur or tibia fracture; 3) Diagnosis with any major cardiovascular or pulmonary disease; 4) Diagnosis with obesity; 5) Diagnosis of lower extremity deep vein thrombosis; 6) Presence of skin lesions or breakdown; 7) Use of electronic implants; 8) Any history of major gastrointestinal problems; 9) difficulty following or responding to commands that would limit the study participation; 10) Currently enrolled in another research study or therapy (from a licensed physical therapist) that is likely to affect participation in this research study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: There will be five participants in each of the three study groups: able-bodied (AB), incomplete spinal cord injury (iSCI), and complete spinal cord injury (cSCI). All participants will be between the ages of 18 and 60 years old. Individuals will be recruited through the Kessler Institute for Rehabilitation System, which includes 3 hospitals and 75 outpatient clinics.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2019-12-09 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Electromyography (EMG) correlates | A single timepoint
  EMG RMS amplitude,
Torque | A single timepoint
  Torque recorded at knee joint using biodex dynamometer

SECONDARY OUTCOMES:
RMSE | single timepoint
  RMSE between EMG feedback vs torque feedback

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided
as per the funding agency guidelines.

REFERENCES:
- [Background] Pilkar R, Yarossi M, Ramanujam A, Rajagopalan V, Bayram MB, Mitchell M, Canton S, Forrest G. Application of Empirical Mode Decomposition Combined With Notch Filtering for Interpretation of Surface Electromyograms During Functional Electrical Stimulation. IEEE Trans Neural Syst Rehabil Eng. 2017 Aug;25(8):1268-1277. doi: 10.1109/TNSRE.2016.2624763. Epub 2016 Nov 3. PMID 27834646
- [Background] Momeni K, Pilkar R, Ravi M, Forrest GF. Isolating Transcutaneous Spinal Cord Stimulation Artifact to Identify Motor Response during Walking. Annu Int Conf IEEE Eng Med Biol Soc. 2021 Nov;2021:6569-6572. doi: 10.1109/EMBC46164.2021.9630099. PMID 34892614